CLINICAL TRIAL: NCT06289790
Title: Analgesic Efficacy of Erector Spinae Plane (ESP) Block vs Intravenous Lignocaine Infusion in Video- Assisted Thoracoscopy (VATS)
Brief Title: Erector Spinae Plane (ESP) Block vs Intravenous Lignocaine Infusion in (VATS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Antoni Okniński, Principal Investigator, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/BW/2023'
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: esp block; lignocaine; Thoracic Surgery, Video-Assisted; erector spinae block
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient and nursing staff will be blinded to the performed intervention. PI and performing anaesthesiologist will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): under general anaesthesia, preoperative ultrasound(USG) guided ESP blockade at Th5, single shot of 30 ml 0,3 % bupivacaine (not exceeding the maximum dose of 2 mg/kg of bupivacaine) with adrenaline 5 µg/ml and dexamethasone 0,15 mg/kg intravenously, post-operative infusion of 0,9% NaCl for 6 hours, infusion rate set as if it were lignocaine 1,5 mg/kg/h
  Interventions: Procedure: Erector Spinae Plane (ESP) block; Drug: Bupivacaine
- Lignocaine infusion group (Active Comparator): pre-induction lignocaine bolus of 1,5 mg/kg i.v. and dexamethasone 0,15 mg/kg intravenously, intraoperative infusion of lignocaine 2 mg/kg i.v., post-operative infusion of lignocaine 1,5 mg/kg i.v. for 6 hours
  Interventions: Drug: Lignocaine

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) block — Erector Spinae Plane (ESP) block with bupivacaine and for pain management in VATS procedure
  Other Names: ESP blockade
  Arms: ESP block group
Drug: Lignocaine — Lignocaine bolus and infusion for pain management in VATS procedure
  Other Names: Lignocaine infusion
  Arms: Lignocaine infusion group
Drug: Bupivacaine — Bupivicaine with adrenaline will be used to perform the ESP block
  Arms: ESP block group

SUMMARY:
The goal of this clinical trial is to compare analgesic efficacy of erector spinae plane (ESP) block vs intravenous lignocaine infusion in video- assisted thoracoscopy (VATS. The main goals are to compare post- operative pain scores and cumulative post- operative opioid doses in both groups

DETAILED DESCRIPTION:
Number of patients: 60 patients enrolled for VATS procedure randomly and evenly assigned to one of the 2 groups.

Randomization: An online tool (Sealed EnvelopeTM[12]) will be used to randomly and evenly assign patients to one of the two groups. Blocks of 4,6,8 will be used and since the blocks assignment will be random as well, the total number of patients can be slightly larger than 60. On the day of the procedure an envelope containing one block of numbers will be opened and numbers from that envelope will be drawn for consecutive patients until the block is finished.

Intervention:

under general anaesthesia, preoperative ultrasound(USG) guided ESP blockade at Th5, single shot of 30 ml 0,3 % bupivacaine (not exceeding the maximum dose of 2 mg/kg of bupivacaine) with adrenaline 5 µg/ml and dexamethasone 0,15 mg/kg intravenously, post-operative infusion of 0,9% NaCl for 6 hours, infusion rate set as if it were lignocaine 1,5 mg/kg/h vs pre-induction lignocaine bolus of 1,5 mg/kg i.v. and dexamethasone 0,15 mg/kg intravenously, intraoperative infusion of lignocaine 2 mg/kg i.v., post-operative infusion of lignocaine 1,5 mg/kg i.v. for 6 hours

Patient and nursing staff will be blinded to the performed intervention.

Primary end- points: 1) pain score (static and dynamic defined as cough effort) on numerical rating score (NRS) 1,3,6,12 hours after surgery (and on discharge from post- anaesthesia care unit [PACU]/after 24 hours- whichever comes sooner) 2) cumulative opioid dose after 12 hours (and on discharge from PACU/after 24 hours- whichever comes sooner)

Secondary end- points: 1) incidence of adverse effects such as: severe hypotension (defined as a 20% drop of either mean arterial pressure (MAP), systolic blood pressure (SBP) or diastolic blood pressure (DBP) compared to baseline measured in the ward prior to surgery)[BP measured at 1,3,6,12 hour and on discharge from PACU or more frequently if needed), nausea and vomiting, priuritis, local anaesthetic systemic toxicity symptoms.

2) intra- operative cumulative opioid dose 3) time to discharge from hospital (max. observation time: 30 days)

ELIGIBILITY:
Inclusion criteria:

* Age >18
* VATS for tumor resection or partial lung resection in emphysema
* Written, informed consent obtained 1 day prior to surgery

Exclusion criteria:

* Lack of consent for ESP blockade
* History of allergy to local anaesthetics
* Other contraindications to ESP blockade
* American Society of Anesthesiologists(ASA) Physical Status Classification value 4 or higher
* VATS for indications other than tumor resection or partial lung resection in emphysema
* Insulin- dependent diabetes mellitus
* More than 1 chest drain post-operatively
* Conversion to thoracotomy
* Chronic opioid use prior to surgery defined as opioid administration for at least 3 months during the last 12 months
* History of alcohol abuse
* Suspected technical difficulties with performing the ESP block (e.g. obesity)
* Inadequate spread of the local anaesthetic during the ESP block
* Cognitive impairment that might cause an inaccurate assessment of pain levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
pain score on numerical rating score | 1,3,6,12 hours after surgery (and on discharge from post- anaesthesia care unit [PACU]/after 24 hours- whichever comes sooner)
  static and dynamic score (defined as cough effort) on numerical rating score (values: 0-10 where the lower number means less pain and a better outcome)
cumulative opioid dose | 12 hours after the end of the surgery (and on discharge from PACU/after 24 hours- whichever comes sooner)
  measured as fentanyl equivalent

SECONDARY OUTCOMES:
incidence of severe hypotension | BP measured at 1,3,6,12 hour and on discharge from PACU or more frequently if needed
  (defined as a 20% drop of either mean arterial pressure (MAP), systolic blood pressure (SBP) or diastolic blood pressure (DBP) compared to baseline measured in the ward prior to surgery
incidence of nausea and vomiting | anytime during post-surgery period until discharge from PACU/after 24 hours- whichever comes sooner
  patients will be monitored for incidence of nausea and vomiting and incidence of those will be noted
incidence of priuritis | anytime during post-surgery period until discharge from PACU/after 24 hours- whichever comes sooner
  patients will be monitored for incidence of priuritis and incidence of it will be noted
incidence of local anaesthetic systemic toxicity symptoms | anytime during post-surgery period until discharge from PACU/after 24 hours- whichever comes sooner
  Patients will be monitored for the following symptoms: limbs numbness, tinnitus, seizures, coma, bradycardia (defined as heart rate below 45 beats per minute), severe ventrical arrhytmias. Incidence of those will be noted.
intra-operative cumulative opioid dose | intra-operative
  measured as fentanyl equivalent
time to discharge from hospital | max. observation time: 30 days
  measured as number of days in the hospital counting from the day of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Okniński, MD, Principal Investigator — National Medical Institute of the Ministry of the Interior and Administration
Locations (1):
- National Medical Institute of the Ministry of the Interior and Administration, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie the results of the publication will be available for researchers upon request and after providing a detailed rationale for obtaining those. All of the data will be deidentified so that the participants will remain anonymous. In order to obtain the data please contact the Principal Investigator at antoni.okninski@cskmswia.gov.pl.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the time of publication. No end date.
Access Criteria: Researchers who provide a sound reason for obtaining the data. Reasearches will need to sign a data access agreement.

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Misiolek H, Zajaczkowska R, Daszkiewicz A, Woron J, Dobrogowski J, Wordliczek J, Owczuk R. Postoperative pain management - 2018 consensus statement of the Section of Regional Anaesthesia and Pain Therapy of the Polish Society of Anaesthesiology and Intensive Therapy, the Polish Society of Regional Anaesthesia and Pain Therapy, the Polish Association for the Study of Pain and the National Consultant in Anaesthesiology and Intensive Therapy. Anaesthesiol Intensive Ther. 2018;50(3):173-199. doi: 10.5603/AIT.2018.0026. PMID 30124229
- [Background] Hou YH, Shi WC, Cai S, Liu H, Zheng Z, Qi FW, Li C, Feng XM, Peng K, Ji FH. Effect of Intravenous Lidocaine on Serum Interleukin-17 After Video-Assisted Thoracic Surgery for Non-Small-Cell Lung Cancer: A Randomized, Double-Blind, Placebo-Controlled Trial. Drug Des Devel Ther. 2021 Aug 3;15:3379-3390. doi: 10.2147/DDDT.S316804. eCollection 2021. PMID 34376972
- [Background] Liu ZJ, Zhang LY, Zheng XG, Shen L, Song KC, Yi J, Huang YG. [Effects of Continuous Intravenous Intraoperative Lidocaine Infusion on Opioids Consumption and Postoperative Recovery in Patients Undergoing Video-assisted Thoracoscopic Lobectomy]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2018 Apr 28;40(2):163-169. doi: 10.3881/j.issn.1000-503X.2018.02.005. Chinese. PMID 29724305
- [Background] Wang L, Sun J, Zhang X, Wang G. The Effect of Lidocaine on Postoperative Quality of Recovery and Lung Protection of Patients Undergoing Thoracoscopic Radical Resection of Lung Cancer. Drug Des Devel Ther. 2021 Apr 7;15:1485-1493. doi: 10.2147/DDDT.S297642. eCollection 2021. PMID 33854301
- [Background] Umari M, Falini S, Segat M, Zuliani M, Crisman M, Comuzzi L, Pagos F, Lovadina S, Lucangelo U. Anesthesia and fast-track in video-assisted thoracic surgery (VATS): from evidence to practice. J Thorac Dis. 2018 Mar;10(Suppl 4):S542-S554. doi: 10.21037/jtd.2017.12.83. PMID 29629201
- [Background] Yao Y, Jiang J, Lin W, Yu Y, Guo Y, Zheng X. Efficacy of systemic lidocaine on postoperative quality of recovery and analgesia after video-assisted thoracic surgery: A randomized controlled trial. J Clin Anesth. 2021 Aug;71:110223. doi: 10.1016/j.jclinane.2021.110223. Epub 2021 Mar 3. PMID 33676296
- [Background] Slovack M, Taylor B, Bryce R, Ong D. Does intravenous lidocaine infusion during video-assisted thoracoscopic surgery reduce postoperative analgesia? A randomized controlled study. Can J Anaesth. 2015 Jun;62(6):676-7. doi: 10.1007/s12630-015-0333-z. Epub 2015 Feb 11. No abstract available. PMID 25670347
- [Background] Gola W, Zając M, Cugowski A. Adiuwanty w blokadach nerwów obwodowych - aktualny stan wiedzy. Anestezjologia Intensywna Terapia. 2020:325-332.
- [Background] Cohen, Edmond. Cohen's Comprehensive Thoracic Anesthesia. Available from: Elsevier eBooks+, Elsevier - OHCE, 2021
- [Background] Sealed Envelope Ltd. 2022. Create a blocked randomisation list. [Online] Available from: https://www.sealedenvelope.com/simple-randomiser/v1/lists